CLINICAL TRIAL: NCT01173705
Title: Genetic and Nutritional Factors Involved in Obesity-related Inflammation and Insulin Resistance
Brief Title: Factors Involved in Obesity-related Inflammation and Insulin Resistance
Status: Terminated | Type: Observational
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Robyn Tamboli, Research Assistant Professor, Vanderbilt University
Organization: Vanderbilt University Medical Center (Other)
Other Study IDs: IRB #100919
Record Dates: First submitted 2010-07-29; First posted 2010-08-02 (Estimated); Last update posted 2017-01-20 (Estimated); Status verified 2017-01

CONDITIONS: Obesity; Insulin Resistance; Inflammation
Keywords: Obesity; Insulin Resistance; Inflammation
MeSH Terms: conditions — Obesity; Insulin Resistance; Inflammation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Whole blood, omentum biopsy, subcutaneous fat biopsy, muscle biopsy (abdominal wall)
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Normal weight: abdominal surgery: Lean individuals undergoing elective abdominal surgery
- Obese: abdominal or bariatic surgery: Obese subjects undergoing elective abdominal or bariatric surgery

SUMMARY:
In this project, we propose to recruit lean and obese subjects with different ethnic background (African Americans and Caucasians) to study the alterations of lipid and carbohydrate metabolism and determine whether these disturbances are linked to genetic, inflammatory, oxidative stress, and/or nutritional factors. Because systemic inflammation and insulin resistance are frequent features of obesity, we postulate that an unbalanced diet with high saturated- and low omega 3-fatty acids is linked to obesity-related inflammation and insulin resistance. We propose to investigate fatty acid metabolism and determine the links between fatty acid composition and oxidative stress in tissues of lean and obese subjects. We propose the following aims:

Specific Aim 1: Evaluate nutrient intake in lean and obese subjects using the standard NHANES Food Questionnaire.

Specific Aim 2: Evaluate the fatty acid composition, including omega-3, in adipose tissue depots, blood monocytes and skeletal muscle, and examine the relationship between omega-3 content and inflammatory and oxidative stress markers.

Specific Aim 3: Compare the effects of omega-3 and saturated FA supplementation on inflammatory and oxidative stress markers in vitro in adipose tissue explants, preadipocytes and monocyte culture.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years of age
* Undergoing elective abdominal or bariatric surgery

Exclusion Criteria:

* Intercurrent infections
* Active cancer diagnosis within 5 years
* Use of medications for diabetes or hyperlipidemia
* Use of glucocorticoids or anti-inflammatory drugs

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Normal weight and obese subjects who are undergoing elective bariatric or abdominal surgery
Sampling Method: Non-Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2011-06; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Examine the relationship between omega-3 content and inflammatory and oxidative stress markers | 5 years
  We will evaluate fatty acid composition in adipose tissues depots, blood monocytes, and skeletal muscle to examine the relationship between omega-e content and inflammatory and oxidative stress markers.

SECONDARY OUTCOMES:
Evaluate nutrient intake | 5 years
  Using the NHANES Food Questionnaire, we will evaluate nutrient intakes of lean and obese individuals
Compare effects of omega-3 and saturated fatty acid supplementation on inflammatory and oxidative stress markers (in vitro) | 5 years
  Compare the effects of omega-3 and saturated FA supplementation on inflammatory and oxidative stress markers in vitro in adipose tissue explants, preadipocytes and monocyte culture.

CONTACTS AND LOCATIONS:
Overall Officials: Robyn Tamboli, PhD, Principal Investigator — Vanderbilt University Medical Center; Naji N Abumrad, MD, Study Chair — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States